CLINICAL TRIAL: NCT06348277
Title: Brief App-based Mood Monitoring and Mindfulness Intervention for First-year College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lawrence University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121119
Record Dates: First submitted 2024-03-20; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Depression, Anxiety; Self-Injurious Behavior
Keywords: mindfulness; rumination; worry
MeSH Terms: conditions — Depression; Anxiety Disorders; Self-Injurious Behavior; Rumination Syndrome | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIndfulness Plus Mood Monitoring (Experimental): Mobile app that involved mood monitoring and brief mindfulness exercises.
  Interventions: Behavioral: Mindfulness plus mood monitoring
- Mood Monitoring Only (Active Comparator): Mobile app that involved only mood monitoring
  Interventions: Behavioral: Mood monitoring
- Assessment only Control (No Intervention): Only completed assessments

INTERVENTIONS:
Behavioral: Mindfulness plus mood monitoring — mobile app that provides guided mindfulness exercises in addition to prompting for mood monitoring three times per day
  Arms: MIndfulness Plus Mood Monitoring
Behavioral: Mood monitoring — mobile app that prompts for mood monitoring three times per day
  Arms: Mood Monitoring Only

SUMMARY:
The investigators examined whether brief, app-based interventions were helpful in alleviating mental health symptoms during the transition to college. In particular, the investigators were interested in whether a brief mobile-app mindfulness intervention combined with mood monitoring was more effective in alleviating first-year students' psychological distress than mood monitoring alone.

DETAILED DESCRIPTION:
The transition to college is associated with worsening mental health symptoms. This study tested whether a brief mobile-app mindfulness intervention combined with mood monitoring was more effective in alleviating first-year students' psychological distress than mood monitoring alone. Participants were 130 first-year students. The investigators randomly assigned 88 students to a mindfulness-plus-mood-monitoring or a mood-monitoring-only group and asked them to use an app 3 times a day for 3 weeks. They, along with an assessment-only control group (n=42), completed self-report questionnaires at baseline, post-intervention, and 6 and 12 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* enrolled first-year student at university

Exclusion Criteria:

* serious suicidal concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | immediately after the intervention
  Beck Depression Inventory; higher scores indicate greater depression
Anxiety Symptoms | immediately after the intervention
  Beck Anxiety Inventory; higher scores indicate greater anxiety
Urges to Self-injure | immediately after the intervention
  Alexian Brothers Urges to Self-Injure scale; higher scores indicate greater urges
Rumination | immediately after the intervention
  Ruminative Response Scale; higher scores indicate higher rumination
Worry | immediately after the intervention
  Penn State Worry Questionnaire; higher scores indicate greater worry

SECONDARY OUTCOMES:
Depressive Symptoms | 6 weeks following the intervention
  Beck Depression Inventory; higher scores indicate greater depression
Depressive Symptoms | 12 weeks following the intervention
  Beck Depression Inventory; higher scores indicate greater depression
Anxiety Symptoms | 6 weeks following the intervention
  Beck Anxiety Inventory; higher scores indicate greater anxiety
Anxiety Symptoms | 12 weeks following the intervention
  Beck Anxiety Inventory; higher scores indicate greater anxiety
Urges to self-injure | 6 weeks following the intervention
  Alexian Brothers Urges to Self-Injure scale; higher scores indicate greater urges
Urges to self-injure | 12 weeks following the intervention
  Alexian Brothers Urges to Self-Injure scale; higher scores indicate greater urges
Rumination | 6 weeks following the intervention
  Ruminative Response Scale; higher scores indicate higher rumination
Rumination | 12 weeks following the intervention
  Ruminative Response Scale; higher scores indicate higher rumination
Worry | 6 weeks following the intervention
  Penn State Worry Questionnaire; higher scores indicate greater worry
Worry | 12 weeks following the intervention
  Penn State Worry Questionnaire; higher scores indicate greater worry

CONTACTS AND LOCATIONS:
Overall Officials: Lori M Hilt, PhD, Principal Investigator — Lawrence University
Locations (1):
- Lawrence University, Appleton, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data available upon request.